CLINICAL TRIAL: NCT05539261
Title: Brain Protection and Neurological Prognosis in Patients With Heart Valve Disease Undergoing Cardiopulmonary Bypass Operation
Brief Title: Research on Neurological Prognosis of Patients Undergoing Heart Valve Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Collaborators: Xi'an Jiaotong University (Other); Yuncheng First Hospital (Unknown)
Responsible Party: Principal Investigator, Qianyan Liu, Principal Investgator, Nanjing University of Traditional Chinese Medicine
Other Study IDs: 82071993
Record Dates: First submitted 2022-09-05; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Heart Valve Diseases; Image
Keywords: Heart Valve Diseases; Cardiopulmonary bypass; MRI Imaging; Neuropsychological assessment
MeSH Terms: conditions — Heart Valve Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HVD: Heart Valve Disease
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale
- HC: Healthy controls
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale

INTERVENTIONS:
Device: magnetic resonance image — Imaging data were collected in a strong magnetic field
Diagnostic Test: Neuropsychological scale — Multi dimensional neuropsychological test

SUMMARY:
The purpose of this study is to clarify the changes of neurocognitive function of patients undergoing cardiac valve disease before and after surgical treatment under cardiopulmonary bypass operation, and to predict the neurological prognosis of such patients through combined imaging technology, so as to improve and avoid the occurrence of postoperative neurological dysfunction in such patients.

DETAILED DESCRIPTION:
This study focuses on brain protection in patients with heart disease. The preoperative brain imaging and consciousness and cognition evaluation results, intraoperative brain monitoring indicators, adverse events of neurological function, brain imaging and consciousness and cognition evaluation results during the postoperative and follow-up periods were recorded. At the same time, serum markers related to perioperative neurological function were obtained to explore the relevant factors affecting neurocognitive function during the perioperative period. The research objectives to investigate the perioperative changes of neurocognitive function in patients undergoing heart valve surgery under cardiopulmonary bypass and the related factors affecting the prognosis of neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-80 years old.
* Accept heart biological valve replacement or heart valvuloplasty.
* More than 6 years of Education.
* At baseline, the score of Mini-mental State Examination (MMSE) scale is more than 23 points

Exclusion Criteria:

* Patients who failed to obtain informed consent.
* Preoperative diagnosis of stroke, epilepsy, history of craniocerebral surgery, cerebrovascular disease, psychosis and rescue patients with cardiopulmonary resuscitation before operation.
* Alcoholism, illiteracy and left-handed.
* There was severe organ hypoperfusion or organ dysfunction before operation, including: preoperative myocardial infarction < 90 days, renal failure or dialysis, severe liver injury, digestive tract ischemia, spinal cord ischemia and iliac artery occlusion.
* There are contraindications to magnetic resonance examination, such as claustrophobia and metal implants in the body.
* Pregnant or lactating women.
* Participating in other clinical studies will affect the main indicators of this study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the patients of HVD group are in-patients and out-patients in the cardiac surgery department from the research center. The subjects of control group are recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of brain volume before and after operation | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of brain volume (mm3) are evaluated by structural 3DT1 weighted MRI. Freesurfer software is used to get the measured value of the volume.
Change of brain function connectivity before and after operation | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of brain functional connectivity intensity are evaluated by rest stage functional MRI. DPABI software based on MATLAB is used to get the measured the matrix value of functional connectivity.

SECONDARY OUTCOMES:
Change of brain evaluate basic cognition before and after operation | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of basic cognition is evaluated by Mini-mental State Examination. The minimum value is 0 , and the maximum value is 30. The higher scores mean a better outcome.
Change of executive functions before and after operation evaluated by Trail-Making Test Part A | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of executive functions are first evaluated by Trail-Making Test Part A test. The minimum value is 0 , and the maximum value is 30. This test has no clear maximum and minimum values. If the test completion time exceeds 79 seconds, it means the outcome is abnormal. The higher scores mean a worse outcome.
Change of executive functions before and after operation evaluated by Digit Symbol Coding score | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of executive functions are second evaluated by Digit Symbol Coding score. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 56.53 ± 20.17. The higher scores mean a better outcome.
Change of working memory before and after operation evaluated by Forward Digit Span | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of working memory is first evaluated by Forward Digit Span. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 7.75±1.47. The higher scores mean a better outcome.
Change of working memory before and after operation evaluated by Backward Digit Span | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of working memory is second evaluated by Backward Digit Span. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 5.36±1.91. The higher scores mean a better outcome.
Change of language ability before and after operation | before operation; 7-10 Days after operation; 1 month; 6-12months
  The change of language ability is evaluated by Chinese Version Verbal Fluency Test. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 19.43±4.81. The higher scores mean a better outcome.
Preliminary judge whether delirium occurs after operation | Witnin 96 hours after operation
  Delirium is preliminary evaluate using confusion assessment method(CAM). The minimum value is 0 , and the maximum value is 4. The higher scores mean a worse outcome.
Fine judge whether delirium occurs after operation | Witnin 96 hours after operation
  Delirium is fine evaluated using Delirium Rating Scale(DRS-R-98). The minimum value is 0 , and the maximum value is 39. The higher scores mean a worse outcome.
Change of plasma marker concentration before and after operation | before operation; immediately after operation; 1,2,3,4 Days after operation
  The change of plasma marker concentration is evaluated by neurofilament light chain(NFL) protein extracted from plasma.
Change of serum marker concentration before and after operation | before operation; immediately after operation; 1,2,3,4 Days after operation
  The change of serum marker concentration is evaluated by inflammatory cytokine.

CONTACTS AND LOCATIONS:
Overall Officials: Nengrui Guo, Principal Investigator — Yuncheng First Hospital
Locations (1):
- Yuncheng First Hospital, Yuncheng, Shanxi, China